CLINICAL TRIAL: NCT00578123
Title: Prospective Assessment of Clinical and Quality of Life Outcomes After Open or Robotic-Assisted Laparoscopic Radical Prostatectomy
Brief Title: Clinical and Quality of Life Outcomes After Open or Robotic-Assisted Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 04-094
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer; Quality of Life
Keywords: Prostate; Cancer; Quality of Life; Questionaires; 04-094
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

ARMS (1):
- 1 Questionnaire (Other): Quality of Life Questionnaires
  Interventions: Behavioral: Quality of Life Questionnaires

INTERVENTIONS:
Behavioral: Quality of Life Questionnaires — Three surveys you will need to complete. We will give you the surveys during your regularly scheduled clinic visits at three, six, and twelve months after surgery. You will NOT be asked to make additional appointments just for the study. You will have the option of completing some of the surveys in an easy to use computer format in the clinic waiting area or on paper.

SUMMARY:
The goal of the study is to look at surgical recovery and quality of life for men who have an open versus robotic-assisted laparoscopic radical prostatectomy (RP). RP is a procedure that removes the prostate gland. We want to see how long it will take you to return to health and strength after surgery. Quality-of-life (QOL) means how you feel about your life and your treatment of prostate cancer. The QOL surveys ask questions about your sexual, urinary and bowel functions. We will also ask questions about your use of health care services, out-of-pocket-spending on medical care and about your return to work, in order to learn about the financial impact of prostate cancer treatment. We hope that the surveys will help show how prostate cancer treatments affect your daily life after surgery.

DETAILED DESCRIPTION:
This study will prospectively assess clinical outcomes in health-related quality of life (HRQOL) in men undergoing open, or robotic-assisted laparoscopic radical prostatectomy. Open radical prostatectomy is a frequently performed treatment for patients with clinically localized (cT1-T2) prostate cancer. The open technique stands as a benchmark against which all other treatments, including new surgical techniques, must be compared. Robotic-assisted and laparoscopic radical prostatectomy is considered an alternative surgical option for clinically localized prostate cancer. While this minimally invasive technique is more frequently being performed in the United States, a detailed comparison of the open and robotic-assisted laparoscopic techniques has not been performed. The relative risks and benefits of these surgical treatment options have not been explored in a contemporary group of patients treated at the same center by surgeons experienced in the open and robotic-assisted laparoscopic techniques. This study will address this deficiency in that follow-up information will be collected prospectively in consecutive patients undergoing open or robotic-assisted laparoscopic radical prostatectomy. While a prospective, randomized trial might be considered a more appropriate methodology to conduct such a comparative study, we have no baseline information, no guidelines to assess robotic-assisted laparoscopic competence, and a lack of skilled robotic-assisted laparoscopic pelvic surgeons to justify a lengthy and expensive trial. We will also collect information on health service utilization and employment during the 12-month postoperative period in order to assess the economic impacts of the different surgical approaches. While results from our proposed study will not necessarily be generalizable to all surgeons and may very well be a comparison of surgeons rather than techniques, the results will provide an initial assessment comparing experts in the open and robotic-assisted laparoscopic techniques. To date, no such comparison has been published. To our knowledge, no other center has expert surgeons in these techniques where such a study would be feasible. Because open techniques have improved dramatically over the past several years, and because the baseline data to be recorded in this proposal is not currently collected, use of historical controls for open radical prostatectomy would be inappropriate.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven adenocarcinoma of the prostate
* Clinical stage T1-T2, NX or N0, Mx or M0
* Life expectancy greater than or equal to 10 years
* Planned radical prostatectomy
* Patients must be able to read and speak English, be free of cognitive impairment, and be reachable by telephone

Exclusion Criteria:

* Prior hormonal therapy for prostate cancer
* Prior pelvic radiation
* Prior chemotherapy for prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 959 (Estimated)
Dates: Start 2005-07; Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
To compare robotic-assisted radical prostatectomy (RALP), and open radical prostatectomy (ORP) with respect to potency function at 1 year, after adjusting for known confounding variables measured at baseline. | 1 year

SECONDARY OUTCOMES:
To evaluate the recovery of continence after RALP or ORP. | 2 years
To evaluate patient convalescence after RALP or ORP. | 2 years
To evaluate operative details. | 2 years
  Including operative time, blood loss, intraoperative fluid requirements, type of anesthesia, number and type of surgical drains, status of the neurovascular bundles including whether or not nerve grafting was performed, incision length, and other ancillary procedures for RALP or ORP
To evaluate inpatient (hospital) details | 2 years
  Including time in the post-anesthesia care unit, hospital convalescence, day of oral intake, day of ambulation, analgesia requirements, daily weights, length of time and output from surgical drains, hemoglobin and creatinine, complications, and length of hospital stay.
To evaluate post-discharge (home) details. | 2 years
  Including analgesic use, return to normal activities/work, time of urinary catheterization, need for catheter replacement, hemoglobin, complications, visit to emergency room or unscheduled clinic visits, and biochemical outcomes (serum PSA levels) following surgery.
To evaluate health service utilization, out-of-pocket spending and changes in employment following RALP or ORP. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org